CLINICAL TRIAL: NCT06972277
Title: The Comparative Effectiveness of Commercial Weight Management Programs in Adults Living With Overweight or Obesity: A Randomized Controlled Trial
Brief Title: A Randomized Controlled Trial Comparing the Efficacy of Commercial Weight Management Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WW International Inc (Industry)
Responsible Party: Principal Investigator, Jamil Alkhaddo, Medical Director, Clinical Development, WW International Inc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: The ACE Study
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Commercial weight management program 1 (Experimental): Participants in this group receive behavioral / lifestyle support from an evidence-based commercial weight management program.
  Interventions: Behavioral: Commercial weight management program
- Commercial weight management program 2 (Experimental): Participants in this group receive behavioral / lifestyle support from an evidence-based commercial weight management program.
  Interventions: Behavioral: Commercial weight management program
- Commercial weight management program 3 (Experimental): Participants in this group receive behavioral / lifestyle support from an evidence-based commercial weight management program.
  Interventions: Behavioral: Commercial weight management program

INTERVENTIONS:
Behavioral: Commercial weight management program — Participants will receive evidence-based behavioral / lifestyle support from a commercial weight management program.

SUMMARY:
The study compares the effectiveness of three commercial weight management programs. The primary outcome is absolute and percentage weight change at 12-weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* BMI ≥27 kg/m²
* Own a bodyweight scale that they can weigh themselves with during the study
* Willing and able to comply with study protocol
* Capable of providing informed consent
* Able to read and write in English
* Willing to be randomized
* Willing to sign a Non Disclosure Agreement

Exclusion Criteria:

* Pregnant, lactating, or plans to become pregnant in the next 6 months
* Previous bariatric surgery or planned bariatric surgery during the study period
* Major surgery within the past 6 months or plans to have surgery during the study period
* Participation in the previous 3 months or current participation in a structured behavioral weight loss program
* Participation in another structured weight loss program during the study period (i.e., the next 3 months)
* Communication needs that would render them unable to understand the study and/or intervention materials
* Current or previous history of anorexia or bulimia nervosa
* Engagement with vomiting or laxative use within the last 28 days with the aim of controlling their shape or weight
* Currently taking anti-obesity medications, planning to take anti-obesity medications in the next 6 months, or previously taken anti-obesity medications in the previous 3 months
* Weight loss of ≥ 5 kg (11 lb) in the previous 6 months
* Self-reported diagnosis of severe depression, bipolar disorder, substance abuse, or psychosis
* Participants who are involved in any other research studies at this time
* Untreated thyroid disease or any changes (type or dose) in thyroid medication in last 6 months
* Chronic/inflammatory gastrointestinal disorders (irritable bowel syndrome is acceptable)
* History of heart problems (e.g., angina, bypass surgery, myocardial infarction, etc.) within previous 6 months
* Diagnosis of type 1 or type 2 diabetes
* Presence of implanted cardiac defibrillator or pacemaker
* History of cancer within past 5 years or current treatment for cancer
* Hospitalization for psychiatric disorders during the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2025-05-14 (Actual); Primary Completion 2026-01-09 (Actual); Study Completion 2026-01-09 (Actual)

PRIMARY OUTCOMES:
Percent body weight lost at 12 weeks | Baseline, 4 weeks, 8 weeks, 12 weeks
  Measurement of weight using a body weight scale
Change in body weight (in kg or pounds) at 12 weeks | Baseline, 4 weeks, 8 weeks, 12 weeks
  Measurement of weight using a body weight scale

SECONDARY OUTCOMES:
Physical Activity and Sedentary Behavior | Baseline, 12 weeks
  Global Physical Activity Questionnaire (GPAQ)
Dietary intake | Baseline, 12 weeks
  Diet ID, powered by Diet Quality Photo Navigation (DQPN®)
Hunger | Baseline, 12 weeks
  Hunger VAS (Visual Analogue Scale)
Impact of Weight on Quality | Baseline, 12 weeks
  Impact of Weight on Quality of Life-Lite (IWQOL-Lite)
Wellbeing | Baseline, 12 weeks
  World Health Organization (WHO-5)
Body appreciation | Baseline, 12 weeks
  Body Appreciation Scale (BAS-2)
Self-Compassion | Baseline, 12 weeks
  Self-Compassion Scale (SCS)
Weight Bias Internalization | Baseline, 12 weeks
  Weight Bias Internalization Scale (WBIS-2F)
Food cravings | Baseline, 12 weeks
  Food Cravings Inventory (FCI-II)

CONTACTS AND LOCATIONS:
Overall Officials: Jamil Alkhaddo, MD, Principal Investigator — WW International Inc
Locations (1):
- WW International, Inc, New York, New York, United States